CLINICAL TRIAL: NCT01006161
Title: Proof-of-Concept and Dose Range-Finding Study of SCH 527123 in Subjects With Severe Asthma
Brief Title: Study of SCH 527123 in Subjects With Severe Asthma (Study P05109AM1)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05109; EUDRACT No.: 2008-004119-36
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — 2-hydroxy-N,N-dimethyl-3-(2-((1-(5-methylfuran-2-yl)propyl)amino)-3,4-dioxocyclobut-1-enylamino)benzamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose SCH 527123 (Experimental)
  Interventions: Drug: SCH 527123
- Medium dose SCH 527123 (Experimental)
  Interventions: Drug: SCH 527123
- High dose SCH 527123 (Experimental)
  Interventions: Drug: SCH 527123
- Placebo (Placebo Comparator)
  Interventions: Drug: SCH 527123

INTERVENTIONS:
Drug: SCH 527123 — Low dose
  Arms: Low dose SCH 527123
Drug: SCH 527123 — Medium dose
  Arms: Medium dose SCH 527123
Drug: SCH 527123 — High dose
  Arms: High dose SCH 527123
Drug: SCH 527123 — Placebo to match SCH 527123
  Arms: Placebo

SUMMARY:
Given the strong inhibition of SCH 527123 on neutrophil migration to sites of inflammation, there is a theoretical reason for its use in patients with severe asthma where neutrophils are thought to play a significant role in the pathophysiology of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have severe asthma, be at least 18 to less than or equal to 70 years of age, of either sex, and any race.

Exclusion Criteria:

* Subject who has been diagnosed with COPD or any other clinically relevant lung disease, other than asthma (eg, cystic fibrosis, pulmonary fibrosis, bronchiectasis).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Severe asthma exacerbations, pulmonary function test data, and a change in symptoms | Measured over the duration of the trial.